CLINICAL TRIAL: NCT06490211
Title: The Research Value of Multi-omics and Multi-modal Information in the Diagnosis and Treatment of Urinary System Tumors
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: S189
Record Dates: First submitted 2024-06-30; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Urinary System Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obtain puncture or surgically removed tumor tissue samples from patients with urinary tract tumors and perform RNA-sequencing, Single-cell RNA-sequence, Spatial Transcriptomics, Proteomics, and Intratumoral Microbiome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients were treated for bladder cancer, kidney cancer, and prostate cancer in Wuhan Union Hospital from January 2024 to January 2026;
2. Aged > 18 years old;
3. Urinalysis, urine exfoliated cells, ultrasound, CT, and MR examinations indicated the above tumors;
4. Tissue biopsy pathological examination confirmed the diagnosis of the above tumors.

Exclusion Criteria:

1. Poor image quality;
2. Incomplete clinical data or loss of follow-up;
3. Presence of another primary malignant tumor other than urinary tract tumor;
4. Unclear pathological diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with urinary system tumors, including kidney cancer, bladder cancer, prostate cancer, etc.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital，Tongji Medical College，Huazhong University of Science and Technology, Wuhan, Hubei, China